CLINICAL TRIAL: NCT06329999
Title: A Prospective, Multicenter, and Exploratory Study of Mitoxantrone Liposomes, Cytarabine and G-CSF Combined With Vineclavone in the Treatment ofRecurrent Adult AML and MDS-EB-2/Elder AML
Brief Title: A Prospective, Multicenter, and Exploratory Study of CMGV in the Treatment of Recurrent Adult AML and MDS-EB-2/Elder AML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Huadong Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Huashan Hospital (Other); Army Medical Center of PLA (Other Government); Sun Yat-sen University (Other); RenJi Hospital (Other); Shanghai Jiading District Central Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); First Hospital of China Medical University (Other); Dalian Municipal Central Hospital (Other); Shanghai Zhongshan Hospital (Other); Shanghai Pudong Hospital (Other); Shanghai Public Health Clinical Center (Other Government); Xuhui Central Hospital, Shanghai (Other); The Affiliated People's Hospital of Ningbo University (Other Government); Taizhou First People's Hospital (Other); Wenzhou People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG-sAML-001
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia
Keywords: Mitoxantrone Hydrochloride Liposomes; Cytarabine; Venetoclax; Recurrent Adult Acute Myeloid Leukemia; MDS-EB-2; Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CMGV regime (Experimental): Mitoxantrone liposomes，Cytarabine，G-CSF，Venetoclax
  Interventions: Drug: CMGV

INTERVENTIONS:
Drug: CMGV — Initial treatment induction therapy: CMG+Vineclavone regimen Mitoxantrone liposomes 15mg/m2, iv, d1; Cytarabine 10mg/m2, H, q12h, d1-7; G-CSF starts at 5ug/kg, H, d0, WBC ≥ 30 × 109/L, stop G-CSF; Vinecla 100mg, 2200mg, 3400mg, d4-10. Every 4 weeks is a cycle, for a total of 2 cycles. For patients with CR/CRI/MLFS/PR in the first cycle, repeat this regimen for consolidation treatment once (the second course of treatment is Vineclavone 400mg d1-7).
  Follow up treatment: Patients who meet the transplantation criteria will undergo hematopoietic stem cell transplantation, while those who do not undergo transplantation will continue to receive CMG+Vineclavone consolidation for 4-6 courses.
  Other Names: CMGV REGIME

SUMMARY:
The goal of this clinical trial] is to evaluate mitoxantrone hydrochloride liposomes, subcutaneous injection of cytarabine and G-CSF combined with Venetoclax (CMG+Ven) in adult secondary acute myeloid leukemia and myelodysplastic syndrome with increased primordial cells type 2(MDS-IB2) or elderly acute myeloid leukemia]. The main questions it aims to answer are:

* Evaluation of the efficacy
* Evaluation of the safety

DETAILED DESCRIPTION:
Mitoxantrone is a traditional anthracycline drug. It exerts anti-tumor effects by interfering with DNA, RNA and inhibiting topoisomerase II. It is a cell cycle non-specific drug ; Mitoxantrone has been used in AML patients. It is widely used in both induction and relapse and refractory treatment stages . At the same time, the literature shows that there is no complete cross-resistance between mitoxantrone and other anthracycline drugs, and it is still effective for patients who have relapsed after previous first-line anthracycline treatment . In addition, the CMG (standard dose cytarabine + mitoxantrone + G-CSF) prestimulation regimen has many applications in China ; a study showed that 16 cases of elderly AML (50% were early in the elderly The CR rate of the CMG regimen for the treatment of secondary AML was 50%, the ORR was 87.4%, and the median OS was 12 months in 2006; a study applied the CMG regimen vs. the conventional dose MA regimen (mitoxantrone + arabinoside Glucoside) in the treatment of elderly AML, the results showed that there was no significant difference in efficacy between the two regimens, but the CMG group had a shorter bone marrow suppression period and less bleeding and infection than the MA group in 2014. Since there is no drug for mitoxantrone in the domestic market for a long period of time, its clinical application is limited. Mitoxantrone Hydrochloride Liposomal Injection is a Class 2 new drug independently developed by CSPC. It will be launched in China in 2022. The approved indications are: those who have received at least first-line standard treatment (including chemotherapy, autologous hematopoietic stem cell transplantation, etc.) For patients with relapsed or refractory peripheral T-cell lymphoma (PTCL), the registration key phase II clinical trial showed good therapeutic effects in relapsed or refractory PTCL and NKTCL, with a confirmed ORR of 41.7%; among them, NKTCL subtype The type has remarkable efficacy, breaking through the limitations of NKTCL's natural resistance to anthracyclines in previous clinical experience. The ORR of single-drug treatment can reach 42.9%.

ELIGIBILITY:
Inclusion Criteria:

* The patient fully understands this study, voluntarily participates and signs an informed consent form (ICF);
* Age: 18-75 years old (including boundary values of 18 and 75);
* Clinically confirmed adult AML and MDS-IB2 (WHO 2022 standard) patients, AML patients meet any of the following criteria:

  1. Treatment related AML
  2. Previously had a history of MDS
  3. Associated with MDS related genes/chromosomal abnormalities
  4. Previously had a history of CMML
  5. Age ≥ 60 years old
  6. Previous history of prodromal MPN, including ET, PV, and MF, with bone marrow fibrosis ≤ grade 2 (according to the 0-3 grade standard)；
* For elderly AML or MDS patients, the comprehensive evaluation should be based on the Fit population: ECOG<3, no major comorbidities, and MMSE and SPPB meet the standards (refer to Appendix 8-11);
* Expected survival time ≥ 3 months;
* Liver and kidney function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal value (ULN) (≤ 5 times the upper limit of normal value for patients with liver infiltration); Total bilirubin ≤ 1.5 times the upper limit of normal value (≤ 3 times the upper limit of normal value for patients with liver infiltration); Serum creatinine ≤ 1.5 times the upper limit of normal value;
* The relevant treatment for MDS (excluding blood transfusion) must be completed 2 weeks before the start of the study treatment; In the case of rapidly proliferative diseases, hydroxyurea is allowed to be used until 24 hours before the start of the study treatment. Before starting the research treatment,Toxicity related to previous MDS treatment must be restored to level 2 or below.

Exclusion Criteria:

The researchers determined that patients who are not suitable to participate in this study. If a patient meets any of the following criteria, they will not be allowed to enter this study:

* The subject's previous history of anti-tumor treatment meets one of the following conditions:

  1. Individuals who have previously received mitoxantrone or mitoxantrone liposomes;
  2. Previously received treatment with doxorubicin or other anthracyclines, with a total cumulative dose of doxorubicin>360mg/m2 (1mg of doxorubicin is equivalent to 2mg of doxorubicin or 0.5mg of doxorubicin);
  3. Within 4 weeks prior to the first use of the study drug or within 5 half-lives of the drug, the patient has received anti-tumor treatment including surgery, chemotherapy, targeted therapy, or participated in other clinical trials and received clinical trial medication;
* Heart function and disease meet one of the following conditions:

  1. Long QTc syndrome or QTc interval>480ms;
  2. Complete left bundle branch block, II or III degree atrioventricular block;
  3. Severe and uncontrolled arrhythmias that require medication treatment;
  4. The New York College of Cardiology in the United States has a classification of ≥ II;
  5. Cardiac ejection fraction (LVEF) below 50%;
  6. A history of myocardial infarction, unstable angina, severe unstable ventricular arrhythmias, or any other arrhythmias requiring treatment, a history of clinically severe pericardial disease, or evidence of acute ischemic or active conduction system abnormalities on electrocardiogram within the 6 months prior to recruitment.
* Patients who have previously or currently suffered from other malignant tumors (except for effectively controlled non melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignant tumors that have not been treated for more than 6 months and have been effectively controlled, as well as patients who have received long-term non chemotherapy treatments such as hormone therapy);
* Uncontrollable systemic diseases (such as infection during the promotion period, uncontrollable hypertension, diabetes, etc.);
* Central nervous system leukemia;
* Secondary AML patients with bone marrow fibrosis ≥ grade 3;
* CML patients with sudden changes;
* Accompanied by a well prognosis chromosome karyotype t (8; 21) (q22; q22.1) RUNX1:: RUNX1T1, inv (16) (p13.1 q22) CBFB: MYH11, as well as acute promyelocytic leukemia;
* Human immunodeficiency virus (HIV) infected individuals (HIV antibody positive);
* Active infection of hepatitis B and hepatitis C (if hepatitis B B surface antigen or core antibody is positive, HBV-DNA will be tested additionally, and if HBV-DNA exceeds 1x103 copies/mL, it will be excluded; if hepatitis C antibody is positive, HCV-RNA will be tested additionally, and if hepatitis C virus RNA exceeds 1x103 copies/mL, it will be excluded);
* Have a known history of immediate or delayed hypersensitivity reactions to similar drugs and excipients in the study drug;
* Accompanied by a history of severe neurological or mental illness;
* The researchers determined that there were patients who were not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
CRc | 1year
  CR (complete remission)+CRi (CR with incomplete recovery of hematological counts)

SECONDARY OUTCOMES:
ORR | 1 year
  Objective Response Rate
OS | 2 year
  Overall Survival
RFS | 2 year
  Relapse-free survival
MRD- | 1 year
  Assessable residual lesion (MRD) conversion rate to negative
Adverse Event | 1 year
  Hematological and non hematological toxicit

CONTACTS AND LOCATIONS:
Overall Officials: sujiang Zhang, Doctor, Principal Investigator — Hematological Depaement, Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No